CLINICAL TRIAL: NCT00885131
Title: Effects of Reward on Learning in the Motor Cortex
Brief Title: Effect of Reward on Learning in Motor Cortex
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Institutes of Health Clinical Center (CC) (NIH); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090124; 09-N-0124
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2013-01-22

CONDITIONS: Healthy
Keywords: Reward Processing; Motor Cortex; HV; Healthy Volunteer

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Magnetic resonance imaging (MRI) uses a strong magnetic field and radio waves to take pictures of the brain. Some MRI studies suggest that this technique reveals brain differences in patients with a nervous system illness when compared to adults without a nervous system illness.

Objectives:

* To study functional changes in the brain that may be observed in people without any nervous system illness.
* To learn more about which areas of the brain are necessary to perform certain tasks, especially learning simple motor sequences and processing rewards.

Eligibility:

* Healthy volunteers between the ages of 18 and 50 who are right-handed and are native English speakers, and who have no medical conditions that would prevent them from undergoing magnetic imaging.
* Volunteers must not have a history of neurological or psychiatric illnesses.
* Female volunteers must not be pregnant.

Design:

* Volunteers will be asked to undergo different types of magnetic imaging, including functional magnetic resonance imaging (fMRI), magnetic resonance spectroscopy (MRS), and/or transcranial magnetic stimulation (TMS), while participating in either a slot machine simulation or a key sequence learning task.
* Volunteers will participate in one of four possible experiments:
* Experiment 1: MRS/TMS and slot machine (3 visits, 3.5 hours in total).
* Experiment 2: MRS/TMS and key sequence (3 visits, 3.5 hours in total).
* Experiment 3: fMRI and slot machine (2 visits, 3 hours in total).
* Experiment 4: fMRI and key sequence (1 visit, 2 hours in total).
* Experiment types:
* Slot machine: A computer game like a slot machine, where the user presses a button to start the game and watches as the three barrels of the machine spin into place.
* Key sequence: Pressing a series of buttons in response to visual cues.
* Volunteers will also be asked to give a small blood sample for genetic testing.
* Volunteers will be paid a small amount of money (approximately $50 $80) during the experiments in compensation for their participation in the study.

DETAILED DESCRIPTION:
Objective: The role of mesencephalic dopamine neurons in reward processing has been established in primates using electrophysiological techniques and in humans using functional neuroimaging. They have rich projections to both the prefrontal and motor cortices where they synapse on interneurons and cortical pyramidal cells, producing primarily inhibition. Though their function is not fully understood, these projections clearly play an important role in motivation and learning. We recently developed a paradigm to detect reward-related signals in the primary motor cortex, using transcranial magnetic stimulation (TMS), and demonstrated increased inhibition in primary motor cortex under conditions of increased reward expectancy. These results suggest that motor learning, which depends critically on the motor cortex, may be influenced by reward, which may take the form of simple performance feedback in humans. This kind of feedback also allows subjects to predict the outcome of actions. Thus, our present objective is to investigate the influence of reward/feedback/prediction on the activity of primary motor cortex during motor learning and in particular during instances of increased reward expectancy. Further, we will examine the role of a brain derived neurotrophic factor (BDNF) single nucleotide polymorphism on motor learning.

Study Population: The population that we will study will be healthy volunteers between the ages of 18-50, without any significant medical history or contraindication to functional magnetic resonance imaging (fMRI).

Design: All experiments will employ within- or between-subjects fMRI and magnetic resonance spectroscopy (MRS) to measure changes in activations of different cortical areas in response to motor learning and reward.

Outcome Measures: The outcome measures will be (a) graded changes in blood oxygen level-dependent (BOLD) in response to motor learning and reward and (b) variations in GABA concentration in response to motor learning and reward, and c) variations in response time in the behavioral performance of a learning task.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-50.
* Right handed.

EXCLUSION CRITERIA:

* Significant neurological or psychiatric history
* Habitual consumption of more than two drinks a day, marijuana more than once a week or any other illicit drug use within the last three months
* Use of medication affecting the DA system, such as phenothiazine antihistamines (promethazine), antiemetics or decongestants within the last month
* Significant abnormality on neurological examination
* Metal in the cranial cavity or eye, pacemaker, implanted pumps or stimulators
* Subjects who participate in any one experiment in this protocol may not participate in another experiment in this protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-04-15; Study Completion 2013-01-22

PRIMARY OUTCOMES:
The outcome measures will be (a) graded changes in blood oxygen level-dependent (BOLD) in response to motor learning and reward and (b) variations in GABA concentration in response to motor learning and reward.

SECONDARY OUTCOMES:
The secondary outcome measures will be variations in response time in the behavioral performance of a learning task.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arancio O, Chao MV. Neurotrophins, synaptic plasticity and dementia. Curr Opin Neurobiol. 2007 Jun;17(3):325-30. doi: 10.1016/j.conb.2007.03.013. Epub 2007 Apr 6. PMID 17419049
- [Background] Ashe J, Lungu OV, Basford AT, Lu X. Cortical control of motor sequences. Curr Opin Neurobiol. 2006 Apr;16(2):213-21. doi: 10.1016/j.conb.2006.03.008. Epub 2006 Mar 24. PMID 16563734
- [Background] Avanzi M, Uber E, Bonfa F. Pathological gambling in two patients on dopamine replacement therapy for Parkinson's disease. Neurol Sci. 2004 Jun;25(2):98-101. doi: 10.1007/s10072-004-0238-z. PMID 15221629